CLINICAL TRIAL: NCT04808999
Title: Phase II Neoadjuvant Study of PD-1 Inhibitor Pembrolizumab in PD-1 Naive Cutaneous Squamous Cell Carcinoma (cSCC)
Brief Title: Neoadjuvant Study of PD-1 Inhibitor Pembrolizumab in PD-1 Naive Cutaneous Squamous Cell Carcinoma (cSCC)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Diwakar Davar (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Diwakar Davar, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 20-300
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Squamous Cell Carcinoma
Keywords: PD-1 inhibitor; neoadjuvant
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab (Experimental): Neoadjuvant Phase: 200 mg IV infusion, every 3 weeks (Day 1 of each 3-week cycle, 2 cycles) Adjuvant Phase: Day 1 of each 3-week cycle, 15 cycles
  Interventions: Drug: Pembrolizumab Injection

INTERVENTIONS:
Drug: Pembrolizumab Injection — 200 mg IV infusion
  Other Names: Keytura

SUMMARY:
This phase II single-arm two-stage neoadjuvant study of pembrolizumab in patients with PD-1 naïve high-risk resectable cutaneous squamous cell carcinoma (cSCC) will be conducted over a 52-week period. The study will include patients who have not undergone surgery to remove disease, to formally evaluate whether both biologically and clinically high-risk disease may benefit from neoadjuvant anti-PD-1 therapy. Response to neoadjuvant anti-PD-1 therapy will be evaluated for association with improved landmark Relapse-free Survival (RFS).

DETAILED DESCRIPTION:
Patients with high-risk resectable cSCC who have yet to undergo definitive surgery will be eligible to enroll. Patients with nodal and/or in-transit relapse including those who have received prior adjuvant RT are eligible to enroll. This trial excludes patients who have received either nivolumab or pembrolizumab or other anti-PD-(L)1 therapy. Suitable patients will be identified pre-operatively. Patients will undergo a 28-day screening evaluation consisting of systemic staging scans, tumor biopsy, and blood studies to confirm suitability. Once enrolled, patients will receive pembrolizumab peri-operatively for 6 weeks (200mg Q3Wq3; 2 cycles) prior to definitive surgery (Neoadjuvant Phase). Following peri-operative therapy, patients will undergo restaging scans and surgical evaluation followed by definitive surgical resection (Surgical Phase). Post-operatively, patients will receive 15 further cycles of pembrolizumab over a 45-week period (200mg q3Q3W) (Adjuvant Phase). In the post-operative period, if patients are deemed eligible for RT, this will be administered concurrently with pembrolizumab. The total duration of pembrolizumab therapy is 1 year (52 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of high-risk localized or locooregional cSCC as defined below may be enrolled in this study.

1. NOTE: Patients are eligible for this trial either at initial presentation for cSCC with locally advanced and/or concurrent regional nodal metastasis; or at the time of recurrence with locally advanced and/or concurrent regional nodal metastasis assuming following criteria are met per the cSCC-specific AJCC UICC 8th edition staging classification

i. T2 and Nx and M0 (tumor >2 cm and ≤4 cm in greatest dimension) OR;

ii. T3 and Nx and M0 (tumor >4 cm or minor bone erosion or perineural invasion or deep invasion) OR;

1. Deep invasion is defined as invasion beyond the subcutaneous fat or >6 mm (as measured from the granular layer of adjacent normal epidermis to the base of the tumor).
2. Perineural invasion is defined as tumor cells within the nerve sheath of a nerve lying deeper than the dermis or measuring 0.1 mm or larger in caliber, or presenting with clinical or radiographic involvement of named nerves without skull base invasion or transgression.

   iii. T4 and Nx and M0 (tumor with gross cortical bone/marrow, skull base invasion and/or skull base foramen invasion if deemed surgically resectable) OR;

   iv. Tx and N1-3 and M0 (if deemed surgically resectable) OR;

   b. NOTE:

   i. If T2, tumors must possess ≥2 NCCN/BWH clinical or pathologic risk factor(s) as stated below.

   ii. NCCN/BWH clinical risk factors:

1. Tumors ≥20 mm on trunk or extremities (excluding pretibia, hands, feet, nail units, and ankles).

2. Tumors ≥10 mm on cheeks, forehead, scalp, neck, or pretibial areas.

iii. NCCN/BWH pathologic risk factors:

1. Poorly defined borders.
2. Recurrent tumors.
3. Neurologic symptoms to suggest perineural invasion.
4. High-risk histologic subtypes including: poorly differentiated tumor, acantholytic (adenoid), adenosquamous, desmoplastic, or metaplastic (carcinosarcomatous) subtypes (as stated in the pathology report or written documentation by Mohs surgeon).
5. Histopathologically documented perineural, lymphatic, or vascular involvement (as stated in the pathology report or written documentation by Mohs surgeon).

   c. NOTE: Tumors of any size on the "mask areas" of the face [central face, eyelids, eyebrows, periorbital nose, lips (cutaneous and vermilion) are not eligible.

   d. NOTE: Tumors of any size on genitalia, hands, and feet may be eligible at the discretion of the treating surgical oncologist.

   e. NOTE: Patients with tumors that arise in the setting of chronic inflammation (Marjolin's ulcer) such as chronic wounds and/or scars are excluded.

   f. NOTE: Determination of surgical resectability must be made before enrollment by the treating surgical oncologist (or ENT surgeon or equivalent).

2. Male participants: A male participant must agree to use a contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.

3. Female participants:

A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

1. Not a woman of childbearing potential (WOCBP)

   OR
2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.

   4. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.

   5. Have at least a single site of measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.

   6. Willing to undergo pre-treatment biopsies.

<!-- -->

1. Prior archival tumor tissue sample are not permitted.
2. Minimum tissue requirements: core (16G or 18G, 6 cores; preferred), punch or excisional biopsy of a tumor lesion that has not been previously irradiated.

   7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.

a. ECOG evaluation should be performed at Screening and repeated on Cycle 1 Day 1.

8. Have adequate organ function, per protocol criteria

Exclusion Criteria:

1. Diagnosis of immunodeficiency, immunosuppression and/or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
3. Prior chemotherapy, targeted small molecule therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
4. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 2-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
6. A WOCBP who has a positive urine pregnancy test at Screening. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
7. Has received a live vaccine within 30 days prior to the first dose of study drug.

   1. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine.
   2. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
8. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 14 days prior to the first dose of study drug.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).

   1. Note: Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
10. Concurrent non-hematologic malignancy other than cSCC within 3 years of data of first planned dose of therapy except for tumors with a negligible risk of metastasis and/or death as defined below:

    a. Adequately treated non-invasive malignancies including but not limited to melanoma in situ (MIS), BCC, CIS of cervix, or DCIS of breast may be enrolled.

    b. Low-risk early stage prostate adenocarcinoma (T1-T2a N0 M0 and Gleason score ≤6 and PSA ≤10 ng/mL) for which the management plan is active surveillance, or prostate adenocarcinoma with biochemical-only recurrence with documented PSA doubling time of > 12 months for which the management plan is active surveillance may be enrolled.

    c. Indolent hematologic malignancies for which the management plan is active surveillance including but not limited to CLL/indolent lymphoma may be enrolled.

    i. Patients with high-risk hematologic malignancies (CML, ALL, AML, Hodgkin's or non- Hodgkin's lymphoma) are excluded even if the management plan is active surveillance.
11. Has known active CNS metastases and/or carcinomatous meningitis.

    a. Note: Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during Screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
12. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
13. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
14. Has an active infection requiring systemic therapy.
15. Has a known history of Human Immunodeficiency Virus (HIV) infection.
16. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) and/or known active Hepatitis C virus (defined as anti-HCV reactive) infection.

    a. Patients with treated Hepatitis B/C with no evidence of active infection may be enrolled.
17. Has a known history of active TB (Bacillus Tuberculosis).
18. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
19. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
20. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the Screening visit through 120 days after the last dose of trial treatment.
21. Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2029-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Diwaker Davar, MD, M.Sc, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.5 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Response
Description: Percentage of patients with either pathologic complete response (pCR) or partial pathologic response (pPR) per Immune-Related Pathologic Response Criteria (immunotherapy-specific pathologic response criteria (irPRC) criteria. Per (irPRC), pCR = 0% residual viable tumor (RVT) remaining in post-therapy specimen (no signs of cancer) in tissue samples removed during surgery, and pPR = >10% but ≤50% RVT remaining in post-therapy specimen in tissue samples removed during surgery.
Time Frame: At time of surgery, up to 6 weeks post-baseline
Population: Treated patients evaluable for pathologic complete response (pCR) at the time of their surgery.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 27
percentage of patients
  pCR | 63.0 [42.4 to 80.6]
  pPR | 7.4 [0.9 to 24.3]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: The median length of time from initiation of study drug(s) until disease relapse (disease progression) as defined by RECIST v1.1, or death. Progressive Disease (PD): ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Time Frame: Up to 60 months
Reporting Status: Not Posted

3. Secondary Outcome: 1-year PRS
Description: The proportion of patients whose disease does not progress/relapse (as defined by RECIST v1.1), or cease to breath at 1 year after the initiation of treatment. Progressive Disease (PD): ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Time Frame: Up to 12 months
Reporting Status: Not Posted

4. Secondary Outcome: 6-month PFS
Description: The proportion of patients whose disease does not progress/relapse (as defined by RECIST v1.1), or cease to breath at 6 months after the initiation of treatment. Progressive Disease (PD): ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Time Frame: Up to 6 months
Reporting Status: Not Posted

5. Secondary Outcome: 2-year PFS
Description: The proportion of patients whose disease does not progress (as defined by RECIST v1.1), or cease to breath at 2 years after the initiation of treatment. Progressive Disease (PD): ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Time Frame: Up to 24 months
Reporting Status: Not Posted

6. Secondary Outcome: 3-year PFS
Description: The proportion of patients whose disease does not progress/relapse (as defined by RECIST v1.1), or cease to breath at 3 years after the initiation of treatment. Progressive Disease (PD): ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Time Frame: Up to 36 months
Reporting Status: Not Posted

7. Secondary Outcome: Overall Survival (OS)
Description: The median length of time from initiation of study treatment that patients remain alive.
Time Frame: Up to 84 months
Reporting Status: Not Posted

8. Secondary Outcome: 1-year OS
Description: The proportion of patients alive at 1 year after the initiation of treatment.
Time Frame: Up to 12 months
Reporting Status: Not Posted

9. Secondary Outcome: 2-year OS
Description: The proportion of patients alive at 2 years after the initiation of treatment.
Time Frame: Up to 24 months
Reporting Status: Not Posted

10. Secondary Outcome: Pathologic Response
Description: Number of patients with response per Immune-Related Pathologic Response Criteria (irPRC) criteria: major pathologic response (<0 to ≤10% RVT); partial pathologic response (<10 to ≤50% RVT).
Time Frame: From start of treatment, up to 24 months
Reporting Status: Not Posted

11. Primary Outcome: Response Assessment Per Immune-Related Pathologic Response Criteria (irPRC)
Description: Number of patients with pathologic complete response (pCR), partial pathologic response (pPR), pathologic non-response (pNR) per Immune-Related Pathologic Response Criteria ((irPRC) criteria. Per (irPRC), pCR = 0% residual viable tumor (RVT) (no signs of cancer), pPR = >10% but ≤50% RVT, or pNR = >50% RVT remaining in post-therapy specimen tissue samples removed during surgery.
Time Frame: At time of surgery
Population: Treated patients evaluable for pathologic complete response (pCR) at the time of their surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 27
Participants
  pCR | 17
  pPR | 2
  pNR | 8

ADVERSE EVENTS:
Time Frame: Adverse Events data collected for a total of approximately 45 months for the study population. Up to approximately 16 months after start of treatment for individuals.
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 6/30
Serious Adverse Events (participants affected / at risk) | 13/30
Other Adverse Events (participants affected / at risk) | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=30)
Cardiac arrest (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 1
Mobitz (type) II atrioventricular block (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 1
GI bleed (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Hepatitis viral (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
Blood bilirubin increased (Investigations) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
metabolic encephalopathy (Nervous system disorders) | 1
nephritis (Renal and urinary disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
skin graft surgery (Surgical and medical procedures) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=30)
Anemia (Blood and lymphatic system disorders) | 17
Eosinophilia (Blood and lymphatic system disorders) | 4
Leukocytosis (Blood and lymphatic system disorders) | 2
Aortic valve disease (Cardiac disorders) | 1
coronary artery disease (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 5
Sinus tachycardia (Cardiac disorders) | 4
ear congestion (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 3
Hypothyroidism (Endocrine disorders) | 5
Eyelid function disorder (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 7
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Oral pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 6
Fatigue (General disorders) | 12
Fever (General disorders) | 1
Flu like symptoms (General disorders) | 1
Gait disturbance (General disorders) | 2
edema - tumor site (General disorders) | 1
erythema - right upper extremity (General disorders) | 1
wound vac at surgical site (General disorders) | 1
Localized edema (General disorders) | 1
Malaise (General disorders) | 1
Pain (General disorders) | 10
immune mediated hepatitis (Immune system disorders) | 1
COVID-19 (Infections and infestations) | 1
aspiration pneumonia (Infections and infestations) | 2
infection - right neck (Infections and infestations) | 1
skin graft to back of head (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Dermatitis radiation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 6
Fracture (Injury, poisoning and procedural complications) | 1
Wound complication (Injury, poisoning and procedural complications) | 3
Activated partial thromboplastin time prolonged (Investigations) | 7
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 8
Blood bilirubin increased (Investigations) | 3
Blood lactate dehydrogenase increased (Investigations) | 15
CPK increased (Investigations) | 4
Cardiac troponin I increased (Investigations) | 2
Creatinine increased (Investigations) | 3
Hemoglobin increased (Investigations) | 2
INR increased (Investigations) | 5
Gout (Investigations) | 1
Lichen-planus-like keratosis right shoulder (Investigations) | 1
Thyroid surgery (Investigations) | 1
multiple actinic keratosis of face and scalp (Investigations) | 1
multiple benign melanocytic nevi (Investigations) | 1
new primary SCC left neck (Investigations) | 1
new primary SCC right mandible (Investigations) | 1
seborrheic keratosis (Investigations) | 1
tumor drainage - clear thick in color (Investigations) | 1
tumor erythema (Investigations) | 1
Lymphocyte count decreased (Investigations) | 9
Lymphocyte count increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 4
Thyroid stimulating hormone increased (Investigations) | 8
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 15
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyperlipidemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 3
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 15
Hypophosphatemia (Metabolism and nutrition disorders) | 7
latent autoimmune diabetes in adults (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
EMZL MALT lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
basal cell carcinoma of left nasal sidewall and left neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
left lateral shoulder SCC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 3
Facial muscle weakness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 5
Paresthesia (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Glucosuria (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 4
Ua Specific Gravity increased (Renal and urinary disorders) | 1
Ua Specific Gravity low (Renal and urinary disorders) | 1
blood urea nitrogen (BUN) increased (Renal and urinary disorders) | 1
specify increased specific gravity (Renal and urinary disorders) | 4
renal cysts (Renal and urinary disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
actinic keratosis (Skin and subcutaneous tissue disorders) | 1
bactrim rash (Skin and subcutaneous tissue disorders) | 1
skin infection (cellulitus) (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1
contrast infiltration (Surgical and medical procedures) | 1
ectropian right lower eyelid/dehiscence of right cheek surgical wound (Surgical and medical procedures) | 1
oral fiberoptic bronchoscopy (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 9
Hypotension (Vascular disorders) | 4
Thromboembolic event (Vascular disorders) | 1
increased specific gravity (Renal and urinary disorders) | 1
Ua Specific Gravity increased (Renal and urinary disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT04808999/Prot_SAP_000.pdf